CLINICAL TRIAL: NCT04347252
Title: Incretin Action in Physiology and Diabetes
Brief Title: Glucagon Regulation of Glucose Metabolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David D'Alessio, M.D. (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, David D'Alessio, M.D., Professor, Division Chief of Endocrinology, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00065698_1; R01DK101991 (NIH)
Record Dates: First submitted 2020-03-31; First posted 2020-04-15 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Insulin Secretion
Keywords: glucagon; GLP-1 receptor; insulin secretion; glucose tolerance
MeSH Terms: interventions — Glucagon; exendin (9-39)

STUDY DESIGN:
Intervention Model Description: Within-subject design with each subject receiving 3 separate single day interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Glucagon at basal glycemia (Experimental): Subjects will present after an overnight fast and at time 0 an infusion of deuterated glucose will be started and continued for the remainder of the 5 hour study (4 mg/kg bolus followed by 0.04 mg/kg/min infusion). Blood will be sampled at 10 minute intervals throughout the study for measurement of substrates and hormones. At time 240 an intravenous infusion of glucagon (10-100 ng.kg.min) will be started and continued for 30 or 60 minutes.
  Interventions: Drug: Glucagon
- Glucagon at hyperglycemia (Experimental): Subjects will present after an overnight fast and at time 0 an infusion of deuterated glucose will be started and continued for the remainder of the 5 hour study (4 mg/kg bolus followed by 0.04 mg/kg/min infusion). Blood will be sampled at 10 minute intervals throughout the study for measurement of substrates and hormones. At time 120 an infusion of 20% glucose, labeled to 2% with deuterated glucose, will be started and adjusted to raise the blood glucose to 8.3 mM for the remainder of the study. At time 240 an intravenous infusion of glucagon (10-100 ng.kg.min) will be started and continued for 30 or 60 minutes.
  Interventions: Drug: Glucagon
- Glucagon at hyperglycemia with GLP-1R blockade (Experimental): Subjects will present after an overnight fast and at time 0 an infusion of deuterated glucose will be started and continued for the remainder of the 5 hour study (4 mg/kg bolus followed by 0.04 mg/kg/min infusion). Blood will be sampled at 10 minute intervals throughout the study for measurement of substrates and hormones. At time 120 an infusion of 20% glucose, labeled to 2% with deuterated glucose, will be started and adjusted to raise the blood glucose to 8.3 mM for the remainder of the study; concurrently exendin-(9-39) will be infused at 750 pmol/kg/min, also for the remaining 180 minutes. At time 240 an intravenous infusion of glucagon (10-100 ng.kg.min) will be started and continued for 30 or 60 minutes.
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon — Intravenous infusion of glucagon at fasting or elevated glycemia. Blockade of the GLP-1 receptor during hyperglycemia with and without glucagon.
  Other Names: exendin-(9-39); hyperglycemia

SUMMARY:
Glucagon is a 30 amino acid peptide hormone that is produced exclusively in alpha-cells of the pancreatic islets. Glucagon binds to a G-protein coupled receptor and activates intracellular signaling by increasing the synthesis of cyclic AMP by adenylate cyclase. The glucagon receptor is most prominently expressed by hepatocytes and the cardinal action of glucagon is to stimulate hepatic glucose output by increasing glycogenolysis and gluconeogenesis. A deep body of literature supports physiologic actions of glucagon to maintain fasting blood glucose and counter-regulate hypoglycemia, and the current view of glucose metabolism is that insulin and glucagon have opposing and mutually balancing effects on glycemia. However, it has long been appreciated that glucagon actually stimulates insulin secretion and islet β-cells express the glucagon receptor and respond to its activation by increasing cAMP.

The most potent stimulus for glucagon release is hypoglycemia and both low glucose per sé, as well as sympathetic nervous system activity are potent activators of the alpha-cell. However, glucagon is also stimulated by elevations of circulating amino acids, including after protein containing meals; this setting is one in which the release of glucagon during a period of elevated glycemia could contribute to postprandial insulin secretion. In fact, we have demonstrated that normal mice injected with glucagon while fasting (BG 75 mg/dl) have a prompt rise in blood glucose, whereas mice given glucagon while feeding (BG 150 mg/dl) increase insulin output 3 fold and have a decrease in glycemia. Moreover, in studies with isolated mouse and human islets we have demonstrated that glucagon stimulates insulin release by activating both the glucagon and GLP-1 receptors. This counter-intuitive observation has been reported by several other groups as well as ours.

In the studies proposed herein we wish to extend our novel observations to humans. The possibility that glucagon acts in the fed state to promote insulin secretion and glucose disposal would change current views of physiology in both healthy and diabetic persons. Moreover, since one of the more promising area of drug development is the creation of peptides that activate multiple receptors (GLP-1 + glucagon, GLP-1 + GIP + glucagon) the results of our studies have potential implications for therapeutics as well.

DETAILED DESCRIPTION:
Subjects will have a screening visit for history, medication usage, and blood work; those who qualify will be offered participation. Subjects will be instructed to consume their usual diet, including at least 200 g carbohydrate, and not to engage in strenuous physical activity for the 3 days prior to a study. After an overnight fast they will present to the CRU at the Stedman Building on the Center for Living campus and have intravenous catheters placed in both forearms, one for infusion of test substances and the other for blood sampling; the sampling arm will be warmed with a heating pad to improve venous blood flow. All studies will start following withdrawal of several basal samples over an extended period:

1. Glucagon infusion in fasting and hyperglycemic subjects: dose finding. Subjects receive graded doses of intravenous glucagon after a 12-14 hour fast. Doses will start at 10 ng/kg/min and be increased to 50 and 100 ng/kg/min at 30 minute intervals. Glucose concentrations will be measured at the bedside using a YSI glucose analyzer. Plasma samples will be collected at 10 minute intervals for assay of insulin, C-peptide, and glucagon. These pilot studies will provide insight into the relative sensitivity of hepatic glucose production (fasting study) and insulin secretion (glucose infusion study) to glucagon. These studies will include up to 10 volunteers each.
2. Effects of glycemia to mediate glucagon-stimulated hepatic glucose production (HGP) and insulin secretion. Following placement of intravenous catheters subjects will have an infusion of saline with a tracer dose of deuterated glucose for the remainder of the 300 minute protocol. [6, 6]2H2 glucose will be started as a 4 mg/kg bolus over 5 minutes followed by a continuous infusion of 0.020-0.4 mg/kg/min. After a 2 hour equilibration period to label the glucose pool, subjects will have A) saline infusion, B) initiation of a hyperglycemic clamp, C) infusion of exendin-(9-39) 750 pmol/kg/min and a hyperglycemic clamp. The clamp will be generated with the infusion of a 20% solution of dextrose enriched to 2% with deuterated glucose. The infusion rate will be started at 30 mg/kg/h and adjusted every 5 minutes until the blood glucose reaches ~150 mg/dl; the infusion will be adjusted thereafter to maintain this level of glycemia. Blood samples will be taken at 10 minute intervals throughout the study to measure: enrichment with [6, 6]2H2 glucose, insulin, glucagon and C-peptide. After 120 minutes of A) tracer alone, B) hyperglycemia, or C) exendin-9 plus hyperglycemia, subjects will receive glucagon as an infusion of 10-100 ng/kg/min for 30 or 60 minutes.

The primary outcome variables from these experiment will be HGP and insulin secretion. The hypothesis to be tested is that glucagon given at fasting glucose levels will cause a rapid rise in HGP and blood glucose (50-150 mg/dl over basal) with a secondary rise of insulin secretion that follows the change in glycemia; and that glucagon given at mild hyperglycemia will promptly stimulate insulin secretion and limit the response of HGP. The protocol and predictions of results are depicted below.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, fasting glucose values ≤ 95 mg/dL or A1c ≤ 5.9%, and no first degree family members with T2DM.

Exclusion Criteria:

* Active infectious, malignant or inflammatory conditions; unstable angina or uncompensated heart failure; pulmonary disorders including COPD and asthma; malabsorptive GI disease; significant hepatic disease; renal insufficiency (eGFR < 60 ml/kg/min); anemia (hematocrit < 34%); pregnancy; and uncontrolled hypertension. Subjects will be excluded if they require daily medications that alter glucose metabolism or GI function (glucocorticoids, psychotropics, narcotics, metoclopramide).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Change in insulin secretion | before and after glucagon administration, up to 1 hour
  Derived from plasma insulin and C-peptide concentrations
hepatic glucose production | before and after glucagon administration, up to 1 hour
  Derived from isotope dilution based on deuterated glucose enrichment

SECONDARY OUTCOMES:
Change in Glucagon concentrations | before and after glucagon administration, up to 1 hour
  Assay of plasma concentrations
Change in Beta-hydroxybutyrate concentrations | before and after glucagon administration, up to 1 hour
  Assay of plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: David D'Alessio, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No